CLINICAL TRIAL: NCT06670235
Title: Effectiveness of Using Upright Versus Lithotomy Birthing Position on Maternal and Newborn Outcomes: A Quasi Experimental Study
Brief Title: Effectiveness of Upright vs. Lithotomy Birthing Position on Maternal and Newborn Outcomes
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hawler Medical University (Other)
Responsible Party: Principal Investigator, WAHIDA ABDULLAH IBRAHIM, Lecturer, Hawler Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Birth Position
Record Dates: First submitted 2024-10-29; First posted 2024-11-01 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Maternal Outcomes; Newborn Complication
Keywords: Upright birthing position; Lithotomy position; Maternal outcomes in childbirth; Newborn outcomes in labor; Birth position comparison; Labor positions and delivery; Effectiveness of birth positions

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Upright Birthing Position Group (Experimental): Participants assigned to the Upright Birthing Position Arm will be encouraged to maintain an upright position during labor and delivery. The upright position includes a squatting. This arm aims to assess the potential benefits of the upright position, such as improved maternal outcomes (e.g., shorter labor duration, reduced need for interventions) and favorable newborn outcomes (e.g., higher Apgar scores, better oxygenation).
  To evaluate the effects of upright positioning on both maternal and newborn outcomes compared to the traditional lithotomy position.
  Interventions: Behavioral: Upright Birthing Position
- Lithotomy Birthing Position (Active Comparator): Participants in the Lithotomy Position Arm will follow the standard hospital practice of delivering in the lithotomy position, where the mother is lying on her back with legs supported in stirrups. This position is widely used in clinical settings and serves as the control arm to compare with the outcomes from the upright birthing position.
  To serve as a control group to provide a comparative measure of maternal and newborn outcomes against the upright birthing position. Outcomes will include maternal comfort, labor duration, intervention requirements, and newborn health indicators.
  Interventions: Behavioral: Lithotomy Birthing Position

INTERVENTIONS:
Behavioral: Upright Birthing Position — This intervention involves encouraging participants to use an upright position during labor and delivery, which may include : squatting, based on their preference and comfort level. Healthcare staff will support the participants in maintaining an upright position throughout labor as much as possible to evaluate its effects on maternal and newborn outcomes.
  Arms: Upright Birthing Position Group
Behavioral: Lithotomy Birthing Position — Participants in this arm will be positioned in the lithotomy position during labor and delivery, which is a common practice in clinical settings. In this position, the mother lies on her back with her legs supported in stirrups. This intervention serves as the control condition to provide a baseline comparison for evaluating outcomes against the upright birthing position.
  Arms: Lithotomy Birthing Position

SUMMARY:
This study investigates the effectiveness of upright versus lithotomy birthing positions on maternal and newborn outcomes. Conducted at the Maternity Teaching Hospital in Erbil City, it employs a quasi-experimental design with 62 women in each group (Intervention and control), comparing outcomes for those encouraged to use upright positions with those in standard lithotomy. Maternal and newborn outcomes will be assessed to provide evidence on how birthing positions impact labor progression, comfort, and delivery results. The findings aim to inform clinical practice and policy, enhancing midwifery care and supporting patient-centered approaches to childbirth. Does the upright birthing position effect on maternal and newborn outcomes? Does the lithotomy birthing position effect on maternal and newborn outcomes? The expected outcomes will decrease the rate of perineal tear , episiotomy , post partum hemorrhage and decreasing the rate of admission to Neonatal Intensive Care Unit (NICU) in newborn.

DETAILED DESCRIPTION:
This quasi-experimental study assesses the impact of upright versus lithotomy birthing positions on maternal and newborn outcomes, aiming to contribute evidence-based recommendations for optimal birthing practices. As childbirth management increasingly prioritizes maternal comfort and positive birth experiences, this research seeks to fill gaps in understanding the clinical efficacy and maternal satisfaction associated with each position.

Conducted at the Maternity Teaching Hospital in Erbil City, the study will recruit 124 pregnant women, divided equally into two groups: one encouraged to adopt upright positions (e.g., squatting) during labor and delivery, and the other following standard lithotomy position practices. A non probability convenience sampling method is employed, with participants meeting specific inclusion criteria such as gestational age, health status, and labor progression factors.

The intervention includes the promotion of upright positions in the experimental group, while both groups receive standardized maternal care. Data on maternal outcomes-such as labor duration, pain levels, and delivery type-and newborn outcomes, including Apgar scores and need for resuscitation, will be collected and analyzed pre- and post-intervention.

The study's goal is to identify whether upright positions correlate with enhanced labor outcomes, reduced intervention rates, and increased maternal satisfaction. Findings are expected to guide clinical guidelines, informing both practitioners and patients on effective, patient-centered birthing positions. This research further aims to influence midwifery education and policy, advocating for practices that align with women's preferences and cultural contexts, ultimately enhancing maternal and neonatal health outcomes through evidence-based childbirth management.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with singleton pregnancies;
* Gestational age ranges from (≥37 to 41+6 weeks);
* Spontaneous labor with no contraindications to upright positions;
* Active phase of first stage labor;
* Age 18-35 years old;
* Normal size fetus with occipito-anterior position;
* Communicate normally and participate voluntary.

Exclusion Criteria:

* Abnormal fetal position (malpresentation) (e,g., persistent occipital-transverse and occipital-posterior position, etc.);
* Risky pregnancy or childbirth complications, such as (preeclampsia, eclampsia, heart disease, cephalic presentation dystocia, antepartum hemorrhage, fetal distress, intra-uterine growth restriction, intra-amniotic infection); and free from any chronic diseases (heart disease, epilepsy, hypertension, diabetes mellitus and renal disease)
* Multiple gestation;
* Cephalopelvic disproportion (CPD);
* Precipitate labor;
* Antenatally diagnosed fetal anomalies;
* Current history of a leg injury, fracture, and deep vein thrombosis.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 124 (Estimated)
Dates: Start 2024-11-10 (Estimated); Primary Completion 2025-10-25 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Maternal Labor Duration | Assessed continuously from the onset of active labor until delivery.
  The total time from the onset of active labor until delivery. Measurement Method: Measured in minutes and seconds recording by using the stopwatch from mobile clock.
Newborn Apgar score | Immediately after delivery , Assessed at 1 minute , 5 minutes and 10 minutes post-delivery
  Apgar score at 1 , 5 and 10 minutes post-delivery, Measurement Method: from 0 to 2, with a maximum total score of 10, (Color, Heart rate, Reflex, Muscle Tone, Breath).
  Total Score Interpretation 7-10: Generally normal; baby is likely to be in good health. 4-6: Intermediate; may need some help with breathing or other care. 0-3: Critical; immediate resuscitative efforts are typically required.

SECONDARY OUTCOMES:
Maternal Perception of Pain and Comfort | Assessed during labor (intervals to be specified, e.g., every 2 hours) and immediately after delivery.
  Maternal self-reported pain level and comfort during labor and delivery, Measurement Method: Visual Analog Scale (VAS) for pain; Likert scale for comfort. A 0 to 10 Likert scale for pain perception provides more granularity and allows patients to more precisely indicate their pain level. Higher scores generally indicate worse outcomes, meaning more intense pain.
  Lower scores indicate better outcomes or less pain. 0 - No Pain
  1 to 3 - Mild Pain: Minimal discomfort . 4 to 6 - Moderate Pain 7 to 9 - Severe Pain 10 - Worst Possible Pain
Postpartum Hemorrhage (PPH) | Estimated immediately following delivery and up to 2 hours postpartum.
  Estimated blood loss during and after delivery. Measurement methods estimation by (measured in milliliters). Measuring blood loss after labor and delivery is critical in assessing maternal health and identifying postpartum hemorrhage (PPH), a leading cause of maternal mortality. Here are common methods for measuring blood loss in a clinical setting: Traditionally, healthcare providers visually assess blood loss by observing and estimating the amount of blood in pads, towels, drapes, and other materials.
  Though commonly used, visual estimation is often inaccurate, tending to underestimate actual blood loss.
  Less than 500 ml is indicated normal and more than 500 ml Indicate severe blood loss or significant intervention needs, signaling a worse outcome and potentially requiring immediate medical action.
Maternal Satisfaction with the Birth Experience | Assessed within the first 2 hours postpartum, typically before hospital discharge.
  Maternal satisfaction with the birth experience is a crucial indicator of quality in maternity care, reflecting the mother's perceptions, emotions, and overall satisfaction with the care received during labor and delivery. A positive birth experience can enhance maternal confidence, strengthen the mother-infant bond, and promote mental health, while a negative experience may contribute to postpartum depression, anxiety, and even trauma.
  Measuring Maternal Satisfaction Maternal satisfaction is often assessed using validated questionnaires, such as the Childbirth Experience Questionnaire (CEQ) by using this items : Highly Dissatisfied, Dissatisfied, Neutral, Satisfied, Highly Satisfied with good outcomes is highly satisfied but bad outcomes is highly dissatisfied.

CONTACTS AND LOCATIONS:
Locations (1):
- Hawler Medical University, Erbil, Kurdistan region 44001, Erbil, Iraq

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhang H, Huang S, Guo X, Zhao N, Lu Y, Chen M, Li Y, Wu J, Huang L, Ma F, Yang Y, Zhang X, Zhou X, Guo R, Cai W. A randomised controlled trial in comparing maternal and neonatal outcomes between hands-and-knees delivery position and supine position in China. Midwifery. 2017 Jul;50:117-124. doi: 10.1016/j.midw.2017.03.022. Epub 2017 Mar 31. PMID 28414983
- [Background] Cook JA, Julious SA, Sones W, Hampson LV, Hewitt C, Berlin JA, Ashby D, Emsley R, Fergusson DA, Walters SJ, Wilson ECF, Maclennan G, Stallard N, Rothwell JC, Bland M, Brown L, Ramsay CR, Cook A, Armstrong D, Altman D, Vale LD. DELTA2 guidance on choosing the target difference and undertaking and reporting the sample size calculation for a randomised controlled trial. Trials. 2018 Nov 5;19(1):606. doi: 10.1186/s13063-018-2884-0. PMID 30400926
- [Background] Fu L, Huang J, Li D, Wang H, Xing L, Wei T, Hou R, Lu H. Effects of Using Sitting Position versus Lithotomy Position during the Second Stage of Labour on Maternal and Neonatal Outcomes and the Childbirth Experience of Chinese Women: A Prospective Cohort Study. Healthcare (Basel). 2023 Nov 20;11(22):2996. doi: 10.3390/healthcare11222996. PMID 37998488
- [Background] Elvander C, Ahlberg M, Thies-Lagergren L, Cnattingius S, Stephansson O. Birth position and obstetric anal sphincter injury: a population-based study of 113 000 spontaneous births. BMC Pregnancy Childbirth. 2015 Oct 9;15:252. doi: 10.1186/s12884-015-0689-7. PMID 26453177
- [Background] Abdolahian S, Ghavi F, Abdollahifard S, Sheikhan F. Effect of dance labor on the management of active phase labor pain & clients' satisfaction: a randomized controlled trial study. Glob J Health Sci. 2014 Mar 30;6(3):219-26. doi: 10.5539/gjhs.v6n3p219. PMID 24762366